CLINICAL TRIAL: NCT03725644
Title: Effectiveness of Floortime Intervention Program for Preschool Children With Autism Spectrum Disorders
Brief Title: Parent Training Program for Preschool Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Ling-Yi Lin, Associate Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-BR-103-065
Record Dates: First submitted 2018-10-26; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- parent-training program (Experimental): Parents in the treatment group received the parent-training program based on the DIR model. The parent-training program encouraged child-initiated activities according to the functional developmental levels. The treatment intensity and duration were the same for both groups including 3-week courses and 11-week home programs. The investigators in this study are two registered pediatric occupational therapists who have at least five years of early intervention experience and had studied the DIR model.
  Interventions: Behavioral: parent-training program
- traditional program (Experimental): Parents in the control group received the traditional program based on the developmental approach. The traditional program provided parent-lead activities that fit child's developmental stage.
  Interventions: Behavioral: traditional program

INTERVENTIONS:
Behavioral: parent-training program — Parents in the treatment group received the training program from the registered pediatric occupational therapist in six hours over three weeks. The occupational therapist provided suggestions and gave feedback. The parents were encouraged to interact with their children for at least 15 hours per week. Between the fourth and 14th weeks, the parents implemented the intervention programs at home and recorded the daily intensity. The occupational therapist met with the parents and children at monthly intervals (the seventh and 11th weeks) at the laboratory to discuss any difficulties they encountered and to practice the child-initiated activities.
  Arms: parent-training program
Behavioral: traditional program — Parents in the control group also conducted a 14-week program. They received six hours of training over three weeks.Between the fourth and 14th weeks, the parents implemented parent-led activities at home and recorded the daily intensity. The parents were encouraged to do activities with their children for at least 15 hours per week. The occupational therapist met with the parents at monthly intervals (the seventh and 11th weeks) at the laboratory to discuss any difficulties they encountered while practicing the parent-led activities.
  Arms: traditional program

SUMMARY:
Previous research has showed that parent-training programs derived from the developmental individual-difference relationship-based model (DIR) could improve the communicative development of children with autism spectrum disorder (ASD). However, the empirical evidence is weak. This study therefore examines whether a DIR-based parent-training program can improve children's adaptive functioning and parents' parenting skills using a rigorous randomized controlled trial design with a dose-matched control group. Forty preschool children with autism spectrum disorder (ASD) and their parents were randomly assigned to the parent-training program group or the traditional program group at the pre-test phase. Both groups received 14-week intervention programs and were assessed using pre- and post-tests. Children's development levels and adaptive functioning were assessed by the Functional Emotional Assessment Scale (FEAS), the Chinese version of Psychoeducational Profile-third edition (CPEP-3), and the Vineland Adaptive Behavior Scales (VABS). In addition, parents' parenting skills were assessed by the FEAS and parenting stress was evaluated by the Parenting Stress Index-Short Form.

DETAILED DESCRIPTION:
Introduction: Preschool children with autism spectrum disorder and their parents face many difficulties in daily lives, including children's adaptive functioning, parenting skills, and parenting stress. Therefore, effective and economical interventions are very important to support them. With appropriate theoretical bases, a parent-training program could be effective, economical, and feasible while the clinical manpower is insufficient. Among current intervention programs, the play concept and the developmental, individual difference, and relationship-based (DIR) model match the philosophy of occupational therapy. Previous research had showed the play- and DIR-based parent-training programs would improve children's communicative development. However, the empirical evidence was still weak due to poor research designs and little research was comprehensively investigated children's adaptive functioning. Moreover, the results of improvement in parenting skills and reduction of parenting stress were not consistent. Aim: This study would implement a dose-matched control group and comprehensive measurements to examine if the play- and DIR-based parent-training program would improve children's adaptive functioning and parents' parenting skills as well as reduce parenting stress. Hypotheses: We hypothesized that the better improvements would show in the parent-training program than those in the traditional program. Method: We recruited 40 preschool children with autism spectrum disorder and their parents and randomly assigned them to either the parent-training program group or the traditional program group after pretest phase. Both of them conducted 14-week intervention programs and were assessed after interventions. Children's development levels and adaptive functioning were assessed by the Functional Emotional Assessment Scale (FEAS), the Chinese version of Psychoeducational Profile-third edition (CPEP-3), and the Vineland Adaptive Behavior Scales (VABS). In addition, parents' parenting skills were assessed by the FEAS and parenting stress was evaluated by the Parenting Stress Index-Short Form.

ELIGIBILITY:
Inclusion Criteria:

1. children with a diagnosis of ASD according to the Diagnostic and Statistics Manual of Mental Disorders - Fifth edition (DSM-5; APA, 2013) by registered pediatric psychiatrists;
2. mild to severe symptoms of ASD according to the Standard Version of Childhood Autism Rating Scale - Second edition (CARS2-ST; Schopler et al., 2010);
3. children aged 36 to 71 months old;
4. children whose primary caregivers (parents who cared for their child for over 15 hours per week - except during sleep time) used Mandarin as their main language;
5. children whose caregivers' educational level were at or above middle school so that they could read manuals and complete the questionnaires.

Exclusion Criteria:

1. children who attended other intensive interventions (e.g., 25 hours per week) or had been diagnosed with additional diseases or disorders;
2. parents who attended other parent-training programs at the same time.

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change Scores of Functional Emotional Assessment Scale | 14 weeks
  The Functional Emotional Assessment Scale (FEAS; Greenspan et al., 2001) is based on six functional developmental levels of the developmental individual-difference relationship-based model and divided into two parts that (1) examine the children's development and (2) assess the parenting skills. All parents in the study were asked to record their parent-child activities as 15-minute videos. All videos were coded using random numbers to hide the research information (e.g. groups and test time). Two videos (pre- and post-test) were reviewed for each child. Using the Chinese version of the Scoring Form translated by Liao et al. (2014; intraclass correlation coefficient = 0.85), each item of the FEAS was rated as 0, 1 or 2. Higher raw scores represent better functions and skills. The total score is summed and ranges from 0 to 80.

SECONDARY OUTCOMES:
Change Scores of Chinese Version of Psychoeducational Profile - Third Edition | 14 weeks
  The performance scale of the Chinese Version of Psychoeducational Profile-3 (Schopler et al., 2005; Heep Hong Society, 2013) comprises six subtests for developmental abilities (cognitive verbal/preverbal, expressive language, receptive language, fine motor, gross motor and visual-motor imitation), which are summed to create communication and motor composites. The score of each item is rated as 0, 1 or 2. All six subtests for developmental abilities can be converted to age-equivalent and composite scores. The communication and motor composites scores range from 0 to 60. The higher the scores are, the better function the children achieve.
Change Scores of Vineland Adaptive Behavior Scales | 14 weeks
  The Vineland Adaptive Behavior Scales (VABS; Sparrow et al., 1984) comprises four domains, that is, communication, daily living skills, socialization and motor skills, for assessing adaptive functioning in children aged 3 to 12 years old. The raw score in each domain and total raw score are converted to an age-equivalent score. The domain scores are also expressed as standard scores with a mean of 100 and standard deviation of 15. The range for each subscale is from 20 to 140. The subscales are summed to compute a total score, ranging from 80 to 560. The higher the scores are, the better adaptive functioning the children achieve.

OTHER OUTCOMES:
Intensity daily logs | 14 weeks
  All parents recorded intensity (intervention hours per day) using the online Google form or paper daily logs so that their compliance with program implementation could be monitored. The parents also recorded the intensity of the regular interventions that the children received.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Yi Lin, Principal Investigator — National Cheng Kung University

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, CSR
Time Frame: starting in January 2023
Access Criteria: Supporting information will be shared to pediatric occupational therapists, researchers, and parents with autism.
URL: https://hdl.handle.net/11296/y642ft

REFERENCES:
- [Result] Liao ST, Hwang YS, Chen YJ, Lee P, Chen SJ, Lin LY. Home-based DIR/Floortime intervention program for preschool children with autism spectrum disorders: preliminary findings. Phys Occup Ther Pediatr. 2014 Nov;34(4):356-67. doi: 10.3109/01942638.2014.918074. Epub 2014 May 27. PMID 24865120